CLINICAL TRIAL: NCT04041947
Title: Assessment of Delirium Frequency and Risk Factors in Pediatric Intensive Care Unit
Brief Title: Delirium Assessment in the Pediatric Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ahmet Yontem, Principal Investigator, Cukurova University
Other Study IDs: CUTF-GOKAEK-82
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Delirium
Keywords: Delirium; Pediatric intensive care
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to show the efficacy of non-pharmacological interventions on preventing pediatric delirium in pediatric intensive care unit

DETAILED DESCRIPTION:
The aim of this study was to show the efficacy of non-pharmacological interventions on preventing pediatric delirium in pediatric intensive care unit. Patients who is followed up for at least 48 hours in pediatric intensive care unit will be included in the study. Parents of patients will be allowed to stay with the patient as long as the conditions of service is appropriate. Parents will provide oral treatments to the patients. Patients will be allowed to spend time with their phone, tablet or toy in accordance with their age. Fellow resident will screen for pediatric delirium each child using the Cornell Assessment of Pediatric Delirium twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Cerebral Performance Category < 5 points
* Patients who stay in PICU >48 hours

Exclusion Criteria:

* Pediatric Cerebral Performance Category > 4 points
* Patients who stay in PICU <48 hours

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children in PICU
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Pediatric delirium frequency | Up to a month
  The effect of non-pharmacological interventions on the prevalence of pediatric delirium

CONTACTS AND LOCATIONS:
Overall Officials: Dinçer Yildizdaş, Professor, Study Chair — Cukurova University Medicine Faculty
Locations (1):
- Cukurova University Medicine Faculty, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided